CLINICAL TRIAL: NCT00124956
Title: Impact of Body Composition on Pharmacokinetics of Doxorubicin in Pediatric Patients
Brief Title: Doxorubicin Pharmacokinetic (PK) Study
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Glaser Pediatric Research Network (Network); Elizabeth Glaser Pediatric AIDS Foundation (Other)
Responsible Party: Principal Investigator, Steven Dubois, Associate Professor of Pediatrics, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-04-050
Record Dates: First submitted 2005-07-07; First posted 2005-07-29 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin

SUMMARY:
This protocol is designed to obtain detailed information on the impact of body composition on the pharmacokinetic behavior of doxorubicin after a single intravenous dose in children 21 years of age or younger. There is no efficacy component. Approximately 9 children will be enrolled at Children's Hospital Boston. The information gained from this study could be very important in developing dosing strategies for doxorubicin in the obese patient population.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be > 1 and ≤ 21 years old.
* All patients must be receiving chemotherapy that includes doxorubicin administered as an infusion of any duration < 24 hours, on either a 1-day or 2-day schedule. This includes bolus and all short infusion schedules.
* All patients or their parents/legal guardians will provide informed consent/assent (as required by law) indicating their awareness of the investigational nature and the risks of this study according to the informed consent process.

Exclusion Criteria:

* Women who are known to be pregnant or lactating
* Patients with significant uncontrolled systemic illness
* Serum glutamic oxaloacetic transaminase (SGOT/AST), serum glutamic pyruvate transaminase (SGPT/ALT) > 3 times the upper limit of normal tested within 14 days prior to infusion
* Bilirubin > the upper limit of normal tested within 14 days prior to infusion
* Patients whose dose of doxorubicin is based on ideal body weight
* Patients who weigh < 12 kilograms at time of screening

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2003-06

PRIMARY OUTCOMES:
To evaluate the relationship between obesity and doxorubicin pharmacokinetics in children

SECONDARY OUTCOMES:
To explore the relationship between PK parameters and the patients' characteristics (age, gender, and ethnicity) and to correlate between PK parameters and DXA data (fat mass, lean tissue mass, and bone mineral content)

CONTACTS AND LOCATIONS:
Overall Officials: Holcombe Grier, MD, Principal Investigator — Dana Farber Cancer Insitute
Locations (1):
- Children's Hospital, Boston, Boston, Massachusetts, United States